CLINICAL TRIAL: NCT01369056
Title: HAART Adherence Among HIV-infected Persons and the Factors Affecting Treatment Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Collaborators: State University of New York - Downstate Medical Center (Other); Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Principal Investigator, Anneli Uusküla, Principal Investigator (Professor of Epidemiology, Department of Public Health), University of Tartu
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MARTH07237
Record Dates: First submitted 2011-06-03; First posted 2011-06-08 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Acute HIV Infection; Acquired Immunodeficiency Syndrome; Medication Adherence
Keywords: antiretroviral therapy, highly active; treatment adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advanced Adherence Counseling (AdvAdh) (Experimental): Please see the Intervention Description section
  Interventions: Behavioral: Advanced Adherence Counseling (AdvAdh)
- Control (No Intervention): Standard of care (including counseling regarding antiretroviral treatment adherence) received by HIV/AIDS patients at the study clinic

INTERVENTIONS:
Behavioral: Advanced Adherence Counseling (AdvAdh) — AdvAdh consists of 3 individual sessions (study months 0, 3, 6) -- patient-centered, non-judgmental, Motivational Interviewing- and theory-based, semi-structured, brief, candid conversations with a trained clinical care nurse using Next Step Counseling (NSC) approach. The intervention targets: 1) accurate information about antiretroviral treatment (ART) (mechanisms of HIV and antiretrovirals) and the development of mental imagery around it; 2) promotion of perceived sense of ease and efficacy in working ART regimen into the context of one's daily life and present life circumstances that may challenge drug use persistence; 3) identification, refinement of skills promoting ease of adhering to one's ART regimen across the diverse and challenges contexts.
  Other Names: Situated Optimal Adherence Estonia (sOAI Estonia)
  Arms: Advanced Adherence Counseling (AdvAdh)

SUMMARY:
The general objective of this study is to evaluate HAART adherence in Estonia and the factors affecting adherence; and the impact of an individual adherence enhancement counselling and treatment monitoring model (Advanced Adherence, AdvAdh), compared to the regular counselling received by HAART patients.

DETAILED DESCRIPTION:
Specific HIV treatment - HAART (Highly Active Antiretroviral Therapy) can suppress HIV replication and consequently preserve the functioning of immune system. HAART therapy is a lifelong treatment with several different concomitantly administered oral medications. According to studies, low adherence to treatment is directly related to patient's knowledge and beliefs about HAART.

Studies have shown the success of different interventions increasing adherence to HAART, but additional studies need to be carried out in order to determine the most effective components of the interventions and the methods most suitable considering the local context, that could be used in everyday work and with limited resources.

The first places to implement the activities directed at improving treatment adherence are medical institutions, i.e. the departments of infectious diseases where HIV-positive individuals receive HAART treatment.

The aims of the study are:

* to determine the rate of adherence to HAART and its associated factors;
* to conduct a small-scale intervention (randomised controlled) study implementing a brief adherence counseling targeting persons receiving HAART.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected;
* ≥18 years of age;
* speak and read either Estonian or Russian;
* receiving or starting a HAART regimen

Exclusion Criteria:

- triple class antiretroviral drug resistance, as determined from a prior resistance test performed in clinical practice, defined according to International Antiviral Society - USA (IAS-USA) interpretive guidelines for genotypic resistance mutations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in HAART adherence level (HIV RNA and CD4 count) | Data analysed at study months 6 and 12
  HAART adherence is monitored and change at month 6 and 12, as compared to baseline is recorded and compared between the AdvAdh intervention and the control group. For assessment of the effects regression analysis is used. Percentage of patients with HIV-1 RNA level <50 copies/mL in the two study groups is measured at baseline and months 6, 12; and changes from the original log10 HIV-1 RNA level and cluster of differentiation four (CD4) count are compared at months 6, 12. Factors related to achieving HIV-1 RNA level of <50 copies/mL and HAART adherence >95% are assessed.

SECONDARY OUTCOMES:
Study subjects retention in study | Data analysed at end of study (month 12)
Change in quality of life of study subjects | Data analysed at study months 6 and 12
  Quality of life of study subjects (SF-10) is measured at baseline and study month 6 and 12 in both study groups. Change from baseline is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Sharma, MD, MSc, Principal Investigator — State University of of New York Downstate Medical Center; Anneli Uusküla, MD, MSc, PhD, Principal Investigator — University of Tartu Department of Public Health
Locations (1):
- Ida-Viru Central Hospital, Kohtla-Järve, Ida-Virumaa, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chesney M. Adherence to HAART regimens. AIDS Patient Care STDS. 2003 Apr;17(4):169-77. doi: 10.1089/108729103321619773. PMID 12737640
- [Background] Lerner BH, Gulick RM, Dubler NN. Rethinking nonadherence: historical perspectives on triple-drug therapy for HIV disease. Ann Intern Med. 1998 Oct 1;129(7):573-8. doi: 10.7326/0003-4819-129-7-199810010-00012. PMID 9758579
- [Background] Altice FL, Springer S, Buitrago M, Hunt DP, Friedland GH. Pilot study to enhance HIV care using needle exchange-based health services for out-of-treatment injecting drug users. J Urban Health. 2003 Sep;80(3):416-27. doi: 10.1093/jurban/jtg053. PMID 12930880
- [Background] Grossberg R, Zhang Y, Gross R. A time-to-prescription-refill measure of antiretroviral adherence predicted changes in viral load in HIV. J Clin Epidemiol. 2004 Oct;57(10):1107-10. doi: 10.1016/j.jclinepi.2004.04.002. PMID 15528063
- [Background] Radloff L. The CES-D scale: a self-report depression scale for research in the general population. Appl Psych Meas. 1977;1:385-401
- [Background] Clayson DJ, Wild DJ, Quarterman P, Duprat-Lomon I, Kubin M, Coons SJ. A comparative review of health-related quality-of-life measures for use in HIV/AIDS clinical trials. Pharmacoeconomics. 2006;24(8):751-65. doi: 10.2165/00019053-200624080-00003. PMID 16898846
- [Background] Simoni JM, Pearson CR, Pantalone DW, Marks G, Crepaz N. Efficacy of interventions in improving highly active antiretroviral therapy adherence and HIV-1 RNA viral load. A meta-analytic review of randomized controlled trials. J Acquir Immune Defic Syndr. 2006 Dec 1;43 Suppl 1(0 1):S23-35. doi: 10.1097/01.qai.0000248342.05438.52. PMID 17133201
- [Background] Malta M, Magnanini MM, Strathdee SA, Bastos FI. Adherence to antiretroviral therapy among HIV-infected drug users: a meta-analysis. AIDS Behav. 2010 Aug;14(4):731-47. doi: 10.1007/s10461-008-9489-7. Epub 2008 Nov 20. PMID 19020970
- [Background] Krusi A, Wood E, Montaner J, Kerr T. Social and structural determinants of HAART access and adherence among injection drug users. Int J Drug Policy. 2010 Jan;21(1):4-9. doi: 10.1016/j.drugpo.2009.08.003. Epub 2009 Sep 10. PMID 19747811
- [Background] Arnsten JH, Demas PA, Farzadegan H, Grant RW, Gourevitch MN, Chang CJ, Buono D, Eckholdt H, Howard AA, Schoenbaum EE. Antiretroviral therapy adherence and viral suppression in HIV-infected drug users: comparison of self-report and electronic monitoring. Clin Infect Dis. 2001 Oct 15;33(8):1417-23. doi: 10.1086/323201. Epub 2001 Sep 5. PMID 11550118
- [Background] Torres-Madriz G, Lerner D, Ruthazer R, Rogers WH, Wilson IB. Work-related barriers and facilitators to antiretroviral therapy adherence in persons living with HIV infection. AIDS Behav. 2011 Oct;15(7):1475-82. doi: 10.1007/s10461-010-9667-2. PMID 20091340
- [Background] Choo PW, Rand CS, Inui TS, Lee ML, Cain E, Cordeiro-Breault M, Canning C, Platt R. Validation of patient reports, automated pharmacy records, and pill counts with electronic monitoring of adherence to antihypertensive therapy. Med Care. 1999 Sep;37(9):846-57. doi: 10.1097/00005650-199909000-00002. PMID 10493464
- [Background] Gross R, Yip B, Lo Re V 3rd, Wood E, Alexander CS, Harrigan PR, Bangsberg DR, Montaner JS, Hogg RS. A simple, dynamic measure of antiretroviral therapy adherence predicts failure to maintain HIV-1 suppression. J Infect Dis. 2006 Oct 15;194(8):1108-14. doi: 10.1086/507680. Epub 2006 Sep 12. PMID 16991085
- [Background] Nachega JB, Hislop M, Dowdy DW, Chaisson RE, Regensberg L, Maartens G. Adherence to nonnucleoside reverse transcriptase inhibitor-based HIV therapy and virologic outcomes. Ann Intern Med. 2007 Apr 17;146(8):564-73. doi: 10.7326/0003-4819-146-8-200704170-00007. PMID 17438315
- [Background] Stone VE. Strategies for optimizing adherence to highly active antiretroviral therapy: lessons from research and clinical practice. Clin Infect Dis. 2001 Sep 15;33(6):865-72. doi: 10.1086/322698. Epub 2001 Aug 13. PMID 11512092
- [Background] Horne R, Buick D, Fisher M, Leake H, Cooper V, Weinman J. Doubts about necessity and concerns about adverse effects: identifying the types of beliefs that are associated with non-adherence to HAART. Int J STD AIDS. 2004 Jan;15(1):38-44. doi: 10.1258/095646204322637245. PMID 14769170
- [Background] Horne R, Cooper V, Gellaitry G, Date HL, Fisher M. Patients' perceptions of highly active antiretroviral therapy in relation to treatment uptake and adherence: the utility of the necessity-concerns framework. J Acquir Immune Defic Syndr. 2007 Jul 1;45(3):334-41. doi: 10.1097/QAI.0b013e31806910e3. PMID 17514019
- [Background] Parsons JT, Golub SA, Rosof E, Holder C. Motivational interviewing and cognitive-behavioral intervention to improve HIV medication adherence among hazardous drinkers: a randomized controlled trial. J Acquir Immune Defic Syndr. 2007 Dec 1;46(4):443-50. doi: 10.1097/qai.0b013e318158a461. PMID 18077833
- [Background] Sorensen JL, Haug NA, Delucchi KL, Gruber V, Kletter E, Batki SL, Tulsky JP, Barnett P, Hall S. Voucher reinforcement improves medication adherence in HIV-positive methadone patients: a randomized trial. Drug Alcohol Depend. 2007 Apr 17;88(1):54-63. doi: 10.1016/j.drugalcdep.2006.09.019. Epub 2006 Oct 23. PMID 17056206
- [Background] Petersen ML, Wang Y, van der Laan MJ, Guzman D, Riley E, Bangsberg DR. Pillbox organizers are associated with improved adherence to HIV antiretroviral therapy and viral suppression: a marginal structural model analysis. Clin Infect Dis. 2007 Oct 1;45(7):908-15. doi: 10.1086/521250. Epub 2007 Aug 20. PMID 17806060
- [Background] Milam J, Richardson JL, McCutchan A, Stoyanoff S, Weiss J, Kemper C, Larsen RA, Hollander H, Weismuller P, Bolan R. Effect of a brief antiretroviral adherence intervention delivered by HIV care providers. J Acquir Immune Defic Syndr. 2005 Nov 1;40(3):356-63. doi: 10.1097/01.qai.0000159710.98960.81. PMID 16249712
- [Background] Reynolds NR, Neidig JL. Characteristics of nausea reported by HIV-infected patients initiating combination antiretroviral regimens. Clin Nurs Res. 2002 Feb;11(1):71-88. doi: 10.1177/105477380201100106. PMID 11845516
- [Background] Wolfe D. Paradoxes in antiretroviral treatment for injecting drug users: access, adherence and structural barriers in Asia and the former Soviet Union. Int J Drug Policy. 2007 Aug;18(4):246-54. doi: 10.1016/j.drugpo.2007.01.012. Epub 2007 Mar 23. PMID 17689372
- [Background] WHO/UNAIDS/UNICEF. Towards universal access: scaling up priority HIV/AIDS interventions in the health sector: progress report, April 2007. http://www.who.int/hiv/mediacentre/universal_access_progress_report_en.pdf
- [Background] Uuskula A, Kals M, Rajaleid K, Abel K, Talu A, Ruutel K, Platt L, Rhodes T, Dehovitz J, Des Jarlais D. High-prevalence and high-estimated incidence of HIV infection among new injecting drug users in Estonia: need for large scale prevention programs. J Public Health (Oxf). 2008 Jun;30(2):119-25. doi: 10.1093/pubmed/fdn014. Epub 2008 Feb 28. PMID 18308743
- [Background] Talu A, Rajaleid K, Abel-Ollo K, Ruutel K, Rahu M, Rhodes T, Platt L, Bobrova N, Uuskula A. HIV infection and risk behaviour of primary fentanyl and amphetamine injectors in Tallinn, Estonia: implications for intervention. Int J Drug Policy. 2010 Jan;21(1):56-63. doi: 10.1016/j.drugpo.2009.02.007. Epub 2009 Apr 22. PMID 19395249
- [Background] Abel-Ollo K, Rahu M, Rajaleid K, Talu A, Ruutel K, Platt L, Bobrova N, Rhodes T, Uuskula A. Knowledge of HIV serostatus and risk behaviour among injecting drug users in Estonia. AIDS Care. 2009 Jul;21(7):851-7. doi: 10.1080/09540120802657522. PMID 20024741
- [Background] Ruutel K, Pisarev H, Loit HM, Uuskula A. Factors influencing quality of life of people living with HIV in Estonia: a cross-sectional survey. J Int AIDS Soc. 2009 Jul 16;12:13. doi: 10.1186/1758-2652-12-13. PMID 19607721
- [Background] Ruutel K, Uuskula A, Minossenko A, Loit HM. Quality of life of people living with HIV and AIDS in Estonia. Cent Eur J Public Health. 2008 Sep;16(3):111-5. doi: 10.21101/cejph.a3461. PMID 18935773
- [Background] Platt L, Bobrova N, Rhodes T, Uuskula A, Parry JV, Ruutel K, Talu A, Abel K, Rajaleid K, Judd A. High HIV prevalence among injecting drug users in Estonia: implications for understanding the risk environment. AIDS. 2006 Oct 24;20(16):2120-3. doi: 10.1097/01.aids.0000247586.23696.20. PMID 17053361
- [Background] Celentano DD, Vlahov D, Cohn S, Shadle VM, Obasanjo O, Moore RD. Self-reported antiretroviral therapy in injection drug users. JAMA. 1998 Aug 12;280(6):544-6. doi: 10.1001/jama.280.6.544. PMID 9707145
- [Background] Lucas GM, Chaisson RE, Moore RD. Highly active antiretroviral therapy in a large urban clinic: risk factors for virologic failure and adverse drug reactions. Ann Intern Med. 1999 Jul 20;131(2):81-7. doi: 10.7326/0003-4819-131-2-199907200-00002. PMID 10419445
- [Background] Shapiro MF, Morton SC, McCaffrey DF, Senterfitt JW, Fleishman JA, Perlman JF, Athey LA, Keesey JW, Goldman DP, Berry SH, Bozzette SA. Variations in the care of HIV-infected adults in the United States: results from the HIV Cost and Services Utilization Study. JAMA. 1999 Jun 23-30;281(24):2305-15. doi: 10.1001/jama.281.24.2305. PMID 10386555
- [Background] Strathdee SA, Palepu A, Cornelisse PG, Yip B, O'Shaughnessy MV, Montaner JS, Schechter MT, Hogg RS. Barriers to use of free antiretroviral therapy in injection drug users. JAMA. 1998 Aug 12;280(6):547-9. doi: 10.1001/jama.280.6.547. PMID 9707146
- [Background] Malow RM, Baker SM, Klimas N, Antoni MH, Schneiderman N, Penedo FJ, Ziskind D, Page B, McMahon R. Adherence to complex combination antiretroviral therapies by HIV-positive drug abusers. Psychiatr Serv. 1998 Aug;49(8):1021-2, 1024. doi: 10.1176/ps.49.8.1021. No abstract available. PMID 9712205
- [Background] Sherer R. Adherence and antiretroviral therapy in injection drug users. JAMA. 1998 Aug 12;280(6):567-8. doi: 10.1001/jama.280.6.567. No abstract available. PMID 9707152
- [Background] Paterson DL, Swindells S, Mohr J, Brester M, Vergis EN, Squier C, Wagener MM, Singh N. Adherence to protease inhibitor therapy and outcomes in patients with HIV infection. Ann Intern Med. 2000 Jul 4;133(1):21-30. doi: 10.7326/0003-4819-133-1-200007040-00004. PMID 10877736
- [Background] Charnaz, K. Constructing Grounded Theory. A Practical Guide Through Qualitative Analysis. London, Sage Publication, 2006.
- [Background] Moller T, Linaker OM. Using brief self-reports and clinician scales to screen for substance use disorders in psychotic patients. Nord J Psychiatry. 2010 Apr;64(2):130-5. doi: 10.3109/08039480903274423. PMID 19883188
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Uuskula A, Kalikova A, Zilmer K, Tammai L, DeHovitz J. The role of injection drug use in the emergence of Human Immunodeficiency Virus infection in Estonia. Int J Infect Dis. 2002 Mar;6(1):23-7. doi: 10.1016/s1201-9712(02)90131-1. PMID 12044297
- See also: Estonian Health Board. Database of infectious diseases statistics. Tallinn, Estonian Health Board, 2010. http://www.terviseamet.ee/nakkushaigused/nakkushaigustesse-haigestumine/hiv-ja-aids.html — http://www.terviseamet.ee/